CLINICAL TRIAL: NCT04966325
Title: A Single-Dose, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Way Crossover Study to Evaluate the Effect of LC350189 on the QTc (Corrected QT) Interval in Healthy Adult Subjects
Brief Title: Thorough QT (TQT) Study to Evaluate the Effect of LC350189 on Cardiac Repolarization in Healthy Male and Female Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LG-GDCL008
Record Dates: First submitted 2021-06-28; First posted 2021-07-19 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Hyperuricemia; Gout; Qt Interval, Variation in
MeSH Terms: conditions — Hyperuricemia; Gout | interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: 4-way cross over
Who Masked: Participant, Investigator
Masking Description: LC350189 and placebo will be administered in a double blind, double-dummy manner. Moxifloxacin will be administered open-label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment T (Therapeutic dose) (Experimental): Single oral dose of 200 mg LC350189 (1 × 200 mg tablet) and 2 × placebo tablets.
  Interventions: Drug: LC350189 200mg
- Treatment ST (Supratherapeutic dose) (Experimental): Single oral dose of 600 mg LC350189 (3 × 200 mg tablets).
  Interventions: Drug: LC350189 600mg
- Treatment P (Placebo) (Placebo Comparator): Single oral dose of 3 × placebo tablets.
  Interventions: Drug: Placebo
- Treatment M (positive control) (Active Comparator): Single oral dose of moxifloxacin 400 mg (1 × 400 mg tablet; open label)
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: LC350189 200mg — Subject will receive an LC350189 200mg as single-dose on Day 1(Period 1) or Day 5(Period 2) or Day 9(Period 3) or Day 13(Period 4)
  Other Names: LC350189 (therapeutic dose)
  Arms: Treatment T (Therapeutic dose)
Drug: Placebo — Subject will receive a Placebo as single-dose on Day 1(Period 1) or Day 5(Period 2) or Day 9(Period 3) or Day 13(Period 4)
  Other Names: Placebo control
  Arms: Treatment P (Placebo)
Drug: Moxifloxacin 400mg — Subject will receive a Moxifloxacin 400mg as single-dose on Day 1(Period 1) or Day 5(Period 2) or Day 9(Period 3) or Day 13(Period 4)
  Other Names: Positive control
  Arms: Treatment M (positive control)
Drug: LC350189 600mg — Subject will receive an LC350189 600mg as single-dose on Day 1(Period 1) or Day 5(Period 2) or Day 9(Period 3) or Day 13(Period 4)
  Other Names: LC350189 (supratherapeutic dose)
  Arms: Treatment ST (Supratherapeutic dose)

SUMMARY:
This is a Phase 1, single-center, randomized, partially double-blind, placebo- and positive controlled, 4-way crossover study to evaluate the effect of a therapeutic and a supratherapeutic dose of LC350189 on the QTcF in healthy male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 to 55 years of age, inclusive, with a body mass index (BMI) 18 to 33 kg/m2, inclusive, at screening.
* The subject is considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
* The subject is able to provide written informed consent and agrees to comply with all protocol requirements.

Exclusion Criteria:

* The subject has a history of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, or angina.
* The subject has a family history of long QT syndrome, Brugada syndrome, or sudden death.
* The subject has a resting HR of <40 bpm or >100 bpm when vital signs are measured at screening or check-in.
* The subject has history or presence of unstable cardiovascular disease, including myocardial infarction, cardiac arrhythmia, or cerebrovascular disease (eg, cerebrovascular accident/stroke or transient ischemic attack).
* The subject has a history of other acute or chronic cardiovascular disease or coronary revascularization surgery (eg, coronary artery bypass graft, percutaneous transluminal coronary angioplasty).
* The subject uses a cardiac pacemaker.
* The subject has a history of any other medical, psychological, or social condition that, in the opinion of the investigator or the medical monitor, would prevent the subject from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern to the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
The placebo-corrected change from baseline in QTcF | Before dosing (Baseline) through 24 hours after the dose on Day 1 in each treatment period
  QTcF will be analyzed using concentration-QT (cQT) modeling

SECONDARY OUTCOMES:
The placebo-corrected change from baseline in HR (heart rate) | Before dosing (Baseline) through 24 hours after the dose on Day 1 in each treatment period
  HR will be evaluated at each postdose time point
The placebo-corrected change from baseline in PR | Before dosing (Baseline) through 24 hours after the dose on Day 1 in each treatment period
  PR will be evaluated at each postdose time point
The placebo-corrected change from baseline in QRS | Before dosing (Baseline) through 24 hours after the dose on Day 1 in each treatment period
  QRS will be evaluated at each postdose time point

CONTACTS AND LOCATIONS:
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined